CLINICAL TRIAL: NCT05148416
Title: Effect of High Intensity Laser in Treatment of Myofascial Trigger Points in Symptomatic Knee Osteoarthritis : A Randomized Single-blinded Controlled Trial
Brief Title: Effect of High Intensity Laser in Treatment of Myofascial Trigger Points in Symptomatic Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant Basiony Ahmed Basiony, physiotherapist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: High Intensity laser knee
Record Dates: First submitted 2021-11-10; First posted 2021-12-08 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Myofascial Trigger Point Pain; Knee Osteoarthritis
MeSH Terms: conditions — Myofascial Pain Syndromes; Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laser group (Experimental): 1. Experimental group (A) the laser group (n=20) which received
  1. high intensity laser therapy(HILT)
  2. knee osteoarthritis conventional exercises program in form of stretching exercises for both vastus medialis and gastrocnemius muscles , ROM exercises for knee flexion and extension , and isometric strengthening exercise of previously mentioned muscles .
  all interventions were done under the supervision of physiotherapist for 30 minutes once a day for 3 days per week during a period of 4 weeks.
  Interventions: Radiation: High intensity laser treatment; Other: knee osteoarthritis conventional exercises program
- the sham group group( B) (Sham Comparator): the Sham group (n= 20) which received
  1. sham HILT
  2. knee osteoarthritis conventional exercises program previously mentioned .
  all interventions were done under the supervision of physiotherapist for 30 minutes once a day for 3 days per week during a period of 4 weeks.
  Interventions: Device: sham HILT.; Other: knee osteoarthritis conventional exercises program

INTERVENTIONS:
Radiation: High intensity laser treatment — 20 patients received high power laser therapy . Zimmer High power laser applied by laser probe perpendicular to and in slight contact with the skin around knee joint , the total energy was delivered to the patient during one session was 1060 j in 3 phases of treatment.
  Other Names: Zimmer High power laser (with 810 and 980 nm and maximal output power of pmax 7 w cw , made in Germany) with serial number : IEC 60825-1:2007
  Arms: Laser group
Device: sham HILT. — 20 patients received placebo laser " sham laser . The same treatment protocol of HILT was given to the sham group, but the laser instrument was switched off during applications. All laser applications were performed by the same physiotherapist.
  Arms: the sham group group( B)
Other: knee osteoarthritis conventional exercises program — knee osteoarthritis conventional exercises program in form of stretching exercises for both vastus medialis and gastrocnemius muscles , ROM exercises for knee flexion and extension , and isometric strengthening exercise of previously mentioned muscles .
  all interventions were done under the supervision of physiotherapist for 30 minutes once a day for 3 days per week during a period of 4 weeks.

SUMMARY:
This study was conducted to investigate the effect of High intensity laser therapy( HILT) on pressure pain threshold, serum cortisol level, passive knee range of motion, and changes of functional disability in patients with active myofascial trigger points(MTrPs) pain associated wit knee osteoarthritis(OA) .

DETAILED DESCRIPTION:
Osteoarthritis (OA) is the most common cause of musculoskeletal pain and disability. It is a chronic degenerative disorder of multifactorial etiology, including acute and/or chronic insults from normal wear and tear, age, obesity and joint injury. The true pathogenesis remains poorly understood. OA is characterized by a degradation of the articular cartilage, resulting in an alteration of its biomechanical properties, which in turn contributes to a focal loss of articular cartilage, loss of joint space, osteophyte formation, focal areas of synovitis, per articular bone remodeling and sub chondral cysts , OA presents with symptoms such as joint pain, stiffness, motion limitations, motor and sensory dysfunction and functional impairments, thus, preventing patients from participating in regular physical activities , The common sites of OA appear on the knees, hands, and hips, whereas knee OA is the most common .

Pain is the most frequent complaint for patients with knee OA to seek medical attention. If left untreated, pain and stiffness can result in a loss of physical function and independence during daily activities. The presence of OA-related knee pain has also been associated with increased risks of physical disability in the community .

Many studies have revealed a discrepancy between patients' reports of pain and their radiographic findings , a plausible option is that the pain originates from the myofascial trigger points (MTrPs) in the surrounding muscles (myofascial pain) and cannot be visualized by imaging.

The term myofascial pain is defined as "the complex of sensory, motor, and autonomic symptoms caused by MTrPs , MTrPs, hyperirritable spots found in the skeletal muscles, are associated with hypersensitive palpable nodules located in a taut band. The spots are painful on compression and may produce characteristic referred pain, referred tenderness, motor dysfunction, and autonomic phenomena.

All studies found a high prevalence of myofascial pain in knee OA patients . study of OA patients, MTrPs were found in all participants, especially in the medial head of the gastrocnemius (92%) and the vastus medialis muscle (67%).

The treatment of MPS includes:

In activation of trigger points, relaxation of taut bands, and breaking the pain-spasm-ischemia-pain cycle. The most widely used treatment methods for MPS are education, exercise, non steroidal anti-inflammatory drugs (NSAIDs), superficial and deep heat, electrotherapy, laser therapy, and local injections.

Laser treatment :

Is non- invasive and painless and can be easily administered in therapy units for a wide range of conditions .

Recently, high-intensity laser therapy (HILT) was introduced to the field of physical therapy. The advantage of HILT over Low level laser therapy(LLLT) is that HILT is able to reach and stimulate the large and/or deep joints that are difficult to reach in LLLT .

The use of HILT has been proven to significantly reduce pain . Previous studies describe the anti-inflammatory, anti-edematous, and analgesic effects of HILT, thus justifying its use in the therapy of pain .

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as II degree bilateral knee OA having active MTrP in vastus medialis and medial head of gastrocnemius muscles and over the calf muscle .
* The patients from both gender aged were ranged from 35 to 55 years.

Exclusion Criteria:

* Reactive synovitis, corticosteroids or hyaluronic acid application during the last six months
* Not indicated and no history of knee joint arthroplastic surgery.
* Malignant tumors and chronic infection.
* Not diagnosed with cushing's syndrome.

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-13 (Actual); Study Completion 2021-04-13 (Actual)

PRIMARY OUTCOMES:
Pain Intensity: change of serum cortisol level was used in many research as pain blood biomarker | The first sample was obtained before the first day of treatment and the second sample was obtained after 4 weeks (1 month) of treatment
  For measuring serum cortisol level, Each patient was drawn two 5 ml blood samples from cubital vein two times.

SECONDARY OUTCOMES:
Pressure pain threshold: The Commander Algometer (JTECH Medical, Midvale, Utah, USA) was used to measure the PPT. | The first measure was obtained before the first day's treatment and the second measure was obtained after 4 weeks of treatment (1 month).
  It's a hand-held tool that uses manual pressure to test pain sensitivity in deeper structures. It's a valid tool that's been widely used. The algometer's tip was positioned on the trigger area, and pressure was increased at a rate of 1 kg per second.
  When the patient expressed discomfort and verified it verbally, the pressure measurement was recorded as kg/cm2, the technique was done three times at 60-second intervals and the average was taken .

OTHER OUTCOMES:
Knee Function: knee injury and osteoarthritis outcome score ( KOOS )Score was used to measure the changes of functional disability. | The first score was taken before the first day's treatment and the second score was taken after 4 weeks of treatment (1 month).
  KOOS is a valid, and reliable questionnaire used for assessing the functional status and quality of life (QoL) of patients with any type of knee injuries and osteoarthritis .It assesses five outcomes: pain , symptoms , activities of daily living , sport and recreation function and knee related quality of life . It is a 42-itemself-reported, joint-specific questionnaire which comprises five subscales: Pain (nine items), Symptoms (seven items), Activities of daily life (ADL) (17 items), Function in Sport and Recreation (Sport/Rec) (five items) and Knee-related quality of life (QoL) (four items). Each item is scored from 0 (no problems) to 4 (extreme problems). For each subscale, the score was normalized to a 0-100 scale with higher scores indicating better status.
Passive Knee range of motion ( ROM): measured by the digital electronic goniometer Halo device through a standard measuring procedure. | The first measure was obtained before the first day's treatment and the second measure was obtained after 4 weeks of treatment (1 month) .
  the Electro Goniometer device is considered as standard, simple, portable, valid and reliable device for measuring joints range of motion

CONTACTS AND LOCATIONS:
Overall Officials: Mona Ebrahim Morsy Elsayed, A. professor, Principal Investigator — Monamorsy_niles@yahoo.com; Shimaa Taha Abou El Kasem, Lecturer, Principal Investigator — dr.shymaelshazly@yahoo.com
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data obtained through this study may be provided to qualified researchers with academic interest in myofascial trigger points pain and application of high intensity laser therapy
Supporting Information: Study Protocol
Time Frame: data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 2 months.
Access Criteria: access to trial Individual participant Data can be requested by qualified researchers .

REFERENCES:
- [Result] Kheshie AR, Alayat MS, Ali MM. High-intensity versus low-level laser therapy in the treatment of patients with knee osteoarthritis: a randomized controlled trial. Lasers Med Sci. 2014 Jul;29(4):1371-6. doi: 10.1007/s10103-014-1529-0. Epub 2014 Feb 1. PMID 24487957
- [Result] Alayat MSM, Aly THA, Elsayed AEM, Fadil ASM. Efficacy of pulsed Nd:YAG laser in the treatment of patients with knee osteoarthritis: a randomized controlled trial. Lasers Med Sci. 2017 Apr;32(3):503-511. doi: 10.1007/s10103-017-2141-x. Epub 2017 Jan 11. PMID 28078503
- [Result] Kim GJ, Choi J, Lee S, Jeon C, Lee K. The effects of high intensity laser therapy on pain and function in patients with knee osteoarthritis. J Phys Ther Sci. 2016 Nov;28(11):3197-3199. doi: 10.1589/jpts.28.3197. Epub 2016 Nov 29. PMID 27942148
- [Result] Yilmaz M, Tarakci D, Tarakci E. Comparison of high-intensity laser therapy and combination of ultrasound treatment and transcutaneous nerve stimulation on cervical pain associated with cervical disc herniation: A randomized trial. Complement Ther Med. 2020 Mar;49:102295. doi: 10.1016/j.ctim.2019.102295. Epub 2020 Jan 3. PMID 32147037
- [Result] Fiore P, Panza F, Cassatella G, Russo A, Frisardi V, Solfrizzi V, Ranieri M, Di Teo L, Santamato A. Short-term effects of high-intensity laser therapy versus ultrasound therapy in the treatment of low back pain: a randomized controlled trial. Eur J Phys Rehabil Med. 2011 Sep;47(3):367-73. Epub 2011 Jun 8. PMID 21654616
- [Result] Stiglic-Rogoznica N, Stamenkovic D, Frlan-Vrgoc L, Avancini-Dobrovic V, Vrbanic TS. Analgesic effect of high intensity laser therapy in knee osteoarthritis. Coll Antropol. 2011 Sep;35 Suppl 2:183-5. PMID 22220431